CLINICAL TRIAL: NCT00047905
Title: The Process of Prenatal Genetic Counseling Using a Simulated Client - A Pilot Study
Brief Title: Pilot Study of the Process of Prenatal Genetic Counseling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030009; 03-HG-0009
Record Dates: First submitted 2002-10-22; First posted 2002-10-23 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2003-04

CONDITIONS: Genetic Counseling
Keywords: Qualitative; Communication Analysis; RIAS; Counseling Models; Videotaping; Prenatal Genetic Counselors; Counseling Process; Video Tape Study; Simulated Clients; Prenatal Genetic Counseling

INTERVENTIONS:
Behavioral: examine the process of prenatal genetic counseling

SUMMARY:
This study will examine the process of prenatal genetic counseling to determine how various client and counselor factors affect the communication process in a counseling session. The specific aims of the study are to:

* Provide information on prenatal genetic counselors' interactions with clients for the basis of a future larger study of the genetic counseling process.
* Determine the average length and the range of length of prenatal genetic counselors' interactions with clients when family history information has already been provided.
* Document on videotape the communication content and interaction dynamics of prenatal genetic counselors interacting with clients in order to:
* Characterize different models of prenatal genetic counseling
* Determine the nature of discussions concerning cystic fibrosis carrier testing within the context of prenatal genetic counseling.
* Examine the impact of prenatal genetic counselors' characteristics (years of experience, training and background, age, clinical setting, anxiety) on the communication content and interaction dynamics of sessions with clients.
* Examine the impact of the presence of a spouse on the communication content and interaction dynamics of prenatal genetic counseling sessions with clients.
* Examine the impact of client verbal emotional cues on the communication content and interaction dynamics of prenatal genetic counseling sessions.

Counselors will be recruited for this study from among practicing prenatal genetic counselors at regional meetings and a national meeting of the National Society of Genetic Counselors. They will perform prenatal genetic counseling sessions with actors in the roles of client and client's spouse. The sessions will be videotaped, and the counselor and actors will fill out questionnaires regarding the characteristics of the counselor and the session.

Counselors may be contacted later to request permission to use segments of their videotaped sessions for creating a video teaching tool for counseling professionals that illustrates different ways to practice the genetic counseling.

DETAILED DESCRIPTION:
The main objective of this pilot study is to provide insight into the process of prenatal genetic counseling that can both inform the practice of prenatal genetic counseling and serve as the springboard to a later, more comprehensive study. The research participants will all be practicing prenatal genetic counselors recruited from regional meetings and a national meeting of the National Society of Genetic Counselors. Participating genetic counselors will be asked to perform a prenatal genetic counseling session with a simulated client (an actor) or simulated clients (actor and actor posing as spouse) presenting with the indication of advanced maternal age. The participating genetic counselors will also be asked to address cystic fibrosis carrier testing within the course of this session. This session will be videotaped. In addition, both the genetic counselor and simulated client will be asked to fill out questionnaires related to characteristics of the counselor and the session itself. The process and content of the genetic counseling communication will be analyzed qualitatively and quantitatively (using Roter Interaction Analysis System). Through these analyses, we hope to both describe the nature of prenatal genetic counseling communication in a relatively large sample and to determine the ways in which a variety of client and counselor factors affect the communication process itself (determined through changes in the RIAS communication codes). In addition, we hope to provide information on the logistics of data collection in order to inform a similar larger study planned to look at the impact of communication on client outcomes.

ELIGIBILITY:
INCLUSION CRITERIA:

Any master's trained genetic counselors attending the 2002 regional meetings and/or a national meeting of the National Society of Genetic Counselors who currently provide prenatal genetic counseling services as part of their professional practices will be included in the study. In addition, any prenatal genetic counselors referred by these individuals, but who did not attend these meetings, will also be eligible to participate.

EXCLUSION CRITERIA:

Genetic counselors who do not practice prenatal counseling training programs will be excluded In addition, master's level students currently in genetic counseling training programs will be excluded from the study because differences in their stages of training and practice development would introduce additional variability into the data set.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Start 2002-10; Study Completion 2003-04

CONTACTS AND LOCATIONS:
Locations (1):
- National Human Genome Research Institute (NHGRI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Bernhardt BA, Biesecker BB, Mastromarino CL. Goals, benefits, and outcomes of genetic counseling: client and genetic counselor assessment. Am J Med Genet. 2000 Sep 18;94(3):189-97. doi: 10.1002/1096-8628(20000918)94:33.0.co;2-e. PMID 10995504
- [Background] Biesecker BB, Peters KF. Process studies in genetic counseling: peering into the black box. Am J Med Genet. 2001 Fall;106(3):191-8. doi: 10.1002/ajmg.10004. PMID 11778979
- [Background] Bernhardt BA, Geller G, Doksum T, Larson SM, Roter D, Holtzman NA. Prenatal genetic testing: content of discussions between obstetric providers and pregnant women. Obstet Gynecol. 1998 May;91(5 Pt 1):648-55. doi: 10.1016/s0029-7844(98)00011-8. PMID 9572205